CLINICAL TRIAL: NCT01950403
Title: Phase I, Randomized, Placebo-Controlled Trial of Linaclotide to Demonstrate Colorectal Bioactivity in Healthy Volunteers
Brief Title: Linaclotide Acetate in Preventing Colorectal Cancer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MAY2012-00-01; NCI-2013-01788 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HHSN2512012000042I; 13-829; MAY2012-00-01 (Other: Mayo Clinic); MAY2012-00-01 (Other: DCP); N01CN00042 (NIH); NCT01912079 (obsolete NCT alias)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer; Healthy, no Evidence of Disease
MeSH Terms: conditions — Colorectal Neoplasms | interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (linaclotide acetate) (Experimental): Participants receive linaclotide acetate PO QD on days 1-7.
  Interventions: Drug: linaclotide acetate; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Participants receive placebo PO QD on days 1-7.
  Interventions: Other: placebo; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: linaclotide acetate — Given PO
  Other Names: Linzess; MD-1100 Acetate; MM-416775
  Arms: Arm I (linaclotide acetate)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial studies the side effects and best dose of linaclotide acetate in preventing colorectal cancer in healthy volunteers. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of linaclotide acetate may prevent colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the pharmacodynamic effect (PD) of linaclotide (linaclotide acetate) (single daily dose x 7 days, stage I cohort dose= 0.870 mg/day) on cyclic guanosine monophosphate (cGMP) levels, based on biopsy samples obtained pre- and post-intervention from the rectum, until an effect is documented.

SECONDARY OBJECTIVES:

I. To confirm the safety and tolerability of linaclotide. II. To assess the pharmacodynamic effect of linaclotide on cGMP levels, analyzed sequentially from the transverse colon to the cecum, if no cGMP effect was observed in the rectum for the primary endpoint.

III. To compare the change in the cGMP levels from baseline to day 7 between all the assigned doses of linaclotide (including placebo), analyzed sequentially from the rectum, transverse colon, and cecum.

IV. If the study proceeds to stage II, the pharmacodynamic effect of linaclotide on cGMP levels will be assessed from day 6 rectal biopsies (un-prepped).

TERTIARY OBJECTIVES:

I. To assess the pharmacodynamic effect of linaclotide on an additional pathway-specific biomarkers relevant to guanylate cyclase C (GCC) signaling (i.e., vasodilator-stimulated phosphoprotein [VASP] phosphorylation) and a marker of general proliferation (Ki67 expression), based on intestinal mucosa biopsy samples obtained by colonoscopy pre- and post-exposure at the anatomical location (rectum, transverse colon, or cecum) in which cGMP is elevated following linaclotide exposure.

OUTLINE: This is a dose-escalation study. Participants are randomized to 1 of 2 treatment arms.

ARM I: Participants receive linaclotide acetate orally (PO) once daily (QD) on days 1-7.

ARM II: Participants receive placebo PO QD on days 1-7.

After completion of treatment, participants are followed up for 21-51 days.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA
* Ability to understand and willingness to sign a written informed consent document and follow study procedures
* Willingness to abstain from grapefruit juice, alcohol, and concomitant medications during study
* Willingness to employ adequate contraception for men and women of childbearing potential; acceptable methods include double barrier methods, intrauterine device (IUD), postmenopausal status documented by serum follicle-stimulating hormone (FSH), and/or documentation of surgical sterilization
* Body mass index < 35 kg/m^2
* Willingness to provide blood and tissue specimens for research purposes
* REGISTRATION INCLUSION CRITERIA
* Participants must have normal organ function and have normal laboratory findings without clinically significant findings
* Satisfactory anesthesia and intestinal preparation, with no findings of advanced adenoma, chronic inflammation, or cancer

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION CRITERIA
* Previous personal history of advanced adenomas (>= 1 cm in maximal diameter, >= 3 in total number, villous morphology, or high-grade dysplasia) or colorectal cancer
* Family history of polyposis syndrome (e.g., familial adenomatous polyposis [FAP], hereditary non-polyposis colorectal cancer [HNPCC]) or colorectal cancer (first degree relatives younger than 60 years old)
* History of gastroparesis
* History of surgery involving the luminal gastrointestinal (GI) tract, including bariatric surgery
* History of celiac disease
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Irritable bowel syndrome, chronic constipation, functional bowel disorders, or colonic motility disorder
* Any malignancy within 3 years of baseline; participants with a history of basal cell or squamous cell skin cancer may be enrolled at the discretion of the investigator
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to linaclotide
* History of difficulty with colonoscopy or abnormal colorectal anatomy
* Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women
* Use of laxatives more than 3 times per week
* Intestinal motility agents, histamine-2 inverse agonists (H-2 blockers), or proton pump inhibitors
* Current use of >= 5 cigarettes/day
* Current use of >= 3 alcoholic drinks/day
* Use anti-platelet agents within two weeks of anticipated colonoscopy
* Use of anti-coagulants within two weeks of anticipated colonoscopy
* History of bleeding/coagulation problems
* Prior intolerance of or contraindications for the use of sedation or anesthetic agents, which would prevent the safe use of sedation for colonoscopy; this includes allergies to eggs and soy products
* Any medical condition judged by the investigator to constitute a risk to safe participation
* REGISTRATION EXCLUSION CRITERIA
* Colonoscopic finding requiring clinical intervention
* Use of any illicit or illegal substances detected by urinary drug screen
* Inadequate pre-intervention bowel preparation, as determined by the study physician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Dose of linaclotide acetate that produces a 60% response rate for cGMP levels in rectal tissue by radioimmunoassay (RIA) | Baseline to 7 days
  The pharmacological effect is measured by the arithmetic difference in mean cGMP levels before and after 7 days of linaclotide acetate in biopsies from the colonoscopy. The mean cGMP value will be calculated based on 2 biopsies from the rectum assessed at each time point. The PD response is measured by the difference in mean cGMP levels after 7 days.

SECONDARY OUTCOMES:
Incidence of adverse events associated with linaclotide acetate assessed using the Common Terminology Criteria for Adverse Events version 4.0 | Up to 51 days
  Summary statistics, frequency tables, and non-parametric tests will be used to describe the distributions of adverse events.
PD effect of linaclotide acetate on cGMP levels from the transverse colon to the cecum | Up to 7 days
Change in cGMP levels between all assigned doses, analyzed sequentially from the rectum, transverse colon, and cecum | Baseline to 7 days
  Summary statistics and nonparametric tests will be used to compare the change in the cGMP levels between the different dose levels of linaclotide acetate and placebo.
PD effect on cGMP levels (Stage II) | Up to 6 days
  Changes in cGMP levels from baseline to day 6 will also be assessed using summary statistics and nonparametric tests.

OTHER OUTCOMES:
PD effect of linaclotide acetate on GCC signaling (i.e., VASP phosphorylation) and general proliferation (Ki67 expression) | Up to 7 days
  Summary statistics, frequency tables, non-parametric tests, and graphical methods will be used to describe the distributions of cGMP levels relative to linaclotide acetate dose levels and biomarkers. Linear and logistic regression models may also be used as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Limburg, Principal Investigator — Mayo Clinic
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States